CLINICAL TRIAL: NCT00022165
Title: Prevention Of Cancer By Intervention With Selenium
Brief Title: Selenium in the Prevention of Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000068791; SURREY-UK-PRECISE; EU-20113
Record Dates: First submitted 2001-08-10; First posted 2004-03-19 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Selenium yeast
  Interventions: Dietary Supplement: selenium
- Selenium yeast 100 micrograms per day (Experimental): 100 micrograms per day
  Interventions: Dietary Supplement: selenium
- Selenium yeast 200 micrograms per day (Experimental): 200 micrograms per day
  Interventions: Dietary Supplement: selenium
- Selenium yeast 300 micrograms per day (Experimental): 300 micrograms per day
  Interventions: Dietary Supplement: selenium

INTERVENTIONS:
Dietary Supplement: selenium

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. Selenium may be effective in preventing cancer. It is not yet known which dose of selenium may be most effective in preventing cancer.

PURPOSE: Randomized pilot study to determine the effectiveness of selenium in preventing cancer in healthy people.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether daily supplementation with selenium significantly reduces total cancer incidence and site-specific cancer incidence in the general population. II. Determine whether this regimen has a beneficial effect on mood.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Participants are stratified according to age (60-64 vs 65-69 vs 70-74). Participants are randomized to one of four arms. Arm I: Participants receive oral placebo once daily. Arm II: Participants receive low-dose oral selenium once daily. Arm III: Participants receive moderate-dose oral selenium once daily. Arm IV: Participants receive high-dose oral selenium once daily. Treatment in all arms continues for up to 2 years in the absence of unacceptable side effects or diagnosis of cancer.

PROJECTED ACCRUAL: A total of 510 patients (170 per stratum) will be accrued for this study within 9-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Healthy men and women No prior diagnosis of cancer except non-melanoma skin cancer

PATIENT CHARACTERISTICS: Age: 60 to 74 Performance status: SWOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No active liver disease No known abnormal liver function Renal: No active kidney disease No known abnormal kidney function Other: HIV negative No diminished mental capacity that would preclude study

PRIOR CONCURRENT THERAPY: No other concurrent selenium supplements (50 ug/day or more)

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 1999-10; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Rayman, DPhil, Study Chair — University of Surrey
Locations (3):
- United Kingdom (3):
  - Hammersmith Hospital, London, England
  - United Kingdom Coordinating Committee on Cancer Research-ABC, Sutton, England
  - University Of Surrey, Guildford